CLINICAL TRIAL: NCT04944212
Title: Prevalence of Vitamin D Deficiency in Pregnant Women and Their Newborns and Their Association With Maternal and Newborns Characteristics
Brief Title: Prevalence of Vitamin D Deficiency in Pregnant Women and Their Fetus in North Jordan
Status: Completed | Type: Observational
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 39/131/2020
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measuring vitamin D serum level using ELIZA — Venous blood will be obtained from pregnant women at the time of admission and from the umbilical cord veins of the newborns immediately after their delivery. The quantitative measurement of 25OHD in serum will be performed using ELIZA.

SUMMARY:
In Jordan, there are few data about the prevalence of hypovitaminosis D in pregnant women and their newborns and factors that affect their levels. Hence, in this study, investigators will :

1. Determine vitamin D levels among newborns born in north Jordan
2. Determine vitamin D levels among pregnant women in north Jordan
3. Study the association between maternal and infants levels of vitamin D
4. Explore the association between maternal and fetal characteristics and maternal and/or fetal vitamin D level
5. Study the effect of low fetal vitamin D on newborn anthropometry
6. Study the effect of maternal vitamin D supplement use during pregnancy in raising cord serum vitamin D levels

DETAILED DESCRIPTION:
This is a cross-sectional study that will be carried out at King Abdullah University Hospital (KAUH). After being approved by the Institutional Review Board (IRB) of KAUH, written informed consents will be obtained from the newborns' mothers.

5 ml of venous blood will be obtained from pregnant women at the time of admission and 3 ml of venous blood will be obtained from the umbilical cord veins of the newborns immediately after their delivery. The quantitative measurement of 25OHD in serum will be performed using ELIZA.

Investigators will determine the means, medians and standard deviations of 25OHD levels among pregnant women and infants in Jordan. In addition, investigators will study the association between maternal and infants levels of 25OHD. Moreover, investigators will investigate the association between maternal level of vitamin D and elective maternal variables including vitamin D supplements during and before pregnancy, sun exposure, age, weight, parity, BMI, & maternal medical problems. In addition, investigators will study the effect of low fetal vitamin D on newborn anthropometry. Finally, investigators will study the effect of maternal vitamin D supplements use during pregnancy in raising cord serum vitamin D levels

ELIGIBILITY:
Inclusion Criteria:

All pregnant women who attend to labour ward with singleton alive pregnancies

Exclusion Criteria:

women with multiple pregnancies or with dead fetuses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with singleton live fetuses who attended to labour ward
Sampling Method: Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Determine maternal and fetal vitamin D level among pregnant women and their newborns in north Jordan | 5 minutes
  Measurement of vitamin D using ELIZA

SECONDARY OUTCOMES:
Study the association between maternal and infants levels of vitamin D. Study factors that affect maternal and fetal vitamin D level | 5 months
  Both are measured using ELIZA

CONTACTS AND LOCATIONS:
Overall Officials: Rawan A Obeidat, Dr, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- King Abdullah University Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided